CLINICAL TRIAL: NCT05858814
Title: A Phase I/II Clinical Trial of RC1012 Injection for the Prevention of Relapse in AML Patients After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: RC1012 Injection (Allo-DNT Cells) for the Prevention of Relapse in AML Patients After Allo-HSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangdong Ruishun Biotech Co., Ltd (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC1012-AML002
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: allo-HSCT; Cell Therapy; AML; off-the-shelf cell product
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC1012 injection (allo-DNT Cells) (Experimental): The trial is divided into two parts: Part A is a dose escalation trial with two dose groups (1.0×10^8 cells/kg, 1.5×10^8 cells/kg at day 0, day 28 and day 56), with 6-12 patients planned to be enrolled. Part B is a dose-expansion randomized controlled trial in which 40-60 patients will receive RC1012 infusions at RP2D dose levels.
  Interventions: Biological: RC1012 injection (allo-DNT cells)

INTERVENTIONS:
Biological: RC1012 injection (allo-DNT cells) — RC1012 injection (allo-DNT cells) are from healthy donors and have been proved to be safe and demonstrated potent cytotoxicity against AML blasts from AML patients in preclinical and preliminary clinical studies. Allo- DNT cells will be collected from healthy donors (NO MHC match needed) and injected into patients. The drug for this study is an off-the-shelf product. Patients DO NOT need to wait for the cell manufacturing.

SUMMARY:
To evaluate the safety and tolerability of RC1012 injection infusion in AML Patients after Allo-HSCT

DETAILED DESCRIPTION:
This study aims to evaluate the safety and tolerability of RC1012 injection infusion in AML Patients after Allo-HSCT.

DNT cells are mature T lymphocytes that comprise 3-10% of T cells in human peripheral blood mononuclear cells (PBMC). Allo-DNT cells from healthy donors have been proved to be safe and demonstrated potent cytotoxicity against AML blasts from AML patients in preclinical and preliminary clinical studies. Allo-DNT cells will be collected from healthy donors (NO MHC match needed) and infused into patients. The drug for this study is an off-the-shelf product. Patients DO NOT need to wait for the cell manufacturing.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the study procedures for follow-up examinations and treatment.
2. Aged 18 to 70 years (including cut-offs), regardless of gender.
3. Subject must be diagnosed with AML according to World Health Organization (WHO) criteria (2016).
4. The subject has received an allogeneic HSCT within 60-100 days, the percentage of malignant primitive cells in the bone marrow is < 5% after HSCT and STR-PCR shows complete donor chimerism.
5. The subject has one of the following high-risk factors for relapse after allo-HSCT: (1) Failure to achieve remission after two courses of induction chemotherapy. (2) Prior history of Myelodysplastic Syndromes (MDS) or Myeloproliferative Neoplasm (MPN). (3) High leukocytes (≥100×10^9/L) combined with Central Nervous System Leukemia (CNSL); (4) Positive Minimal Residual Disease (MRD) before HSCT; (5) Non-remission or disease progression prior to HSCT; (6) Subject with cytogenetic high-risk factors (except that who can be treated with targeted drugs).
6. The subject has recovered from the toxicity of the prior treatment, i.e., CTCAE toxicity grade <2 (unless the abnormality is tumor-related).
7. ECOG score 0 to 1.
8. With appropriate organ function:

   * Glutathione aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN);
   * Glutamic aminotransferase (ALT) ≤ 3 times ULN;
   * Total bilirubin ≤ 1.5 times ULN, unless the patient has documented Gilbert syndrome. Patients with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included;
   * Serum creatinine ≤ 1.5 times ULN or a creatinine clearance ≥ 60 ml/min;
   * Hemoglobin ≥ 80 g/L or hemoglobin maintained at that level following transfusion;
   * International Normalized Ratio (INR) ≤ 1.5 times ULN and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN;
   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
   * A platelet count ≥ 50 x 10^9/L or a platelet count maintained at that level following a platelet transfusion;
   * Left ventricular ejection fraction (LVEF) ≥ 45%.
9. Female patients with childbearing potential should have a negative pregnancy test during the screening period. Any male and female patients of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female patients without childbearing potential (meeting at least 1 of the following criteria) is described below.

   * Have undergone a hysterectomy or bilateral oophorectomy;
   * Medically recognized as ovarian failure;
   * Medically recognized as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause).

Exclusion Criteria:

1. Subject is confirmed to have morphological relapse of leukemia or positive MRD after allo-HSCT.
2. Subject with extramedullary infiltration of leukemia.
3. Suffer from other malignancies within 5 years prior to screening, except adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, post-radical thyroid cancer, and post-radical ductal carcinoma in situ.
4. Has severe respiratory disease (previous or combined history of severe interstitial lung disease, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm).
5. A previous history of a definite neurological or psychiatric disorder, including epilepsy or dementia.
6. Evidence of active central nervous system invasion or cranial neuropathy.
7. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titration assay not within the normal reference range, positive hepatitis C virus (HCV) antibody and peripheral blood HCV RNA ,positive for human immunodeficiency virus (HIV), or positive for cytomegalovirus (CMV) DNA, or positive syphilis test.
8. Subject who is allergic to the excipients of RC1012 injection or other drugs recommended in the study protocol (e.g., tolimumab, etc.).
9. Serious cardiac disease, including but not limited to severe arrhythmia, unstable angina, massive heart attack, New York Heart Association class III or IV cardiac insufficiency, refractory hypertension.
10. Persons who have previously received an organ transplant or are preparing to receive an organ transplant (except for HSCT).
11. Subject who has received other maintenance therapy drugs after HSCT or who wish to receive other maintenance therapy.
12. Subject with the presence of acute GvHD of degree III to IV or extensive chronic GvHD.
13. Active neurological autoimmune or inflammatory diseases (e.g. Guillain-Barre Syndrome (GBS), Amyotrophic lateral sclerosis (ALS)).
14. Clinically significant active cerebrovascular disease (e.g. cerebral oedema, Posterior Reversible Encephalopathy Syndrome (PRES)).
15. Subject with a life expectancy of less than 3 months.
16. Subject has been involved in other clinical studies within 3 months prior to screening.
17. Subject , in the judgement of the investigator and/or clinical criteria, is contraindicated to any study procedure or have other medical conditions that may place them at unacceptable risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-05-27 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of allo-DNT Cell Therapy for AML subjects after Allo-HSCT
Maximum Tolerated Dose (MTD) | Up to 28 days
  MTD was the highest dose for DLT in ≤1/6 subjects
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 2 years
  The peak concentration of allo-DNT cells amplified in the peripheral blood (Cmax, detected by Flow Cytometry).
Pharmacokinetics (PK) indicator (AUC) | Up to 2 years
  Allo-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by Flow Cytometry).
Pharmacokinetics (PK) indicator (Tmax) | Up to 2 years
  Allo-DNT cells blood concentrations will be measured at different time points to evaluate the peak time (Tmax) in peripheral blood. Tmax is defined as the time to reach the highest concentration (Tmax, detected by Flow Cytometry).
Pharmacokinetics (PK) indicator (T1/2) | Up to 2 years
  Allo-DNT cells blood concentrations will be measured at different time points to evaluate the elimination half-life in hours (T1/2). T1/2 is defined as the time point when the concentration of allo-DNT reaches half of maximum in a patient's peripheral blood (T1/2, detected by Flow Cytometry).
Recurrence rate at 6 months | Up to 6 months
  Record the proportion of patients with recurrence in the study.
Relapse-free survival (RFS) | Up to 2 years
  Relapse-free survival is the time from study enrollment until documented disease relapse, or death from any cause.
GvHD-free and relapse-free survival (GRFS) | Up to 2 years
  GRFS is the time from study enrollment until documented disease relapse, or death, or GvHD occur from any cause.
2-year overall survival | Up to 2 years
  From the date of entry into the clinical study until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, MD, PhD, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- The First Hospital of the University of Science and Technology of China, Hefei, Anhui, China